CLINICAL TRIAL: NCT02832167
Title: An Open Label Phase 2 Multi-cohort Trial of Nivolumab in Advanced or Metastatic Malignancies
Brief Title: An Open Label Investigational Immuno-therapy Trial of Nivolumab in Cancers That Are Advanced or Have Spread
Acronym: CheckMate 627
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-627; 2016-000461-23 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2016-07-08; First posted 2016-07-14 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental)
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo

SUMMARY:
The purpose of this study is to determine whether nivolumab is an effective treatment for cancer that has advanced or has spread. Various tumor types may be eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced or metastatic malignancy
* Received standard of care treatment for primary malignancy and standard of care treatment for relapsed cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Prior treatment with an antiPD1, antiPDL1, antiPDL2, antiCD137, or antiCTLA4 antibody, or any other antibody or drug specifically targeting Tcell co-stimulation or checkpoint pathways.
* Subjects previously treated with investigational anticancer therapies less than 6 weeks prior to the first dose of Nivolumab
* Subjects with an active, known, or suspected autoimmune disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (45):
- United States (39):
  - Arizona Oncology Associates, PC, Tucson, Arizona
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Jude Hospital Yorba Linda, Fullerton, California
  - LACN, Los Angeles, California
  - UCLA Main Campus - University California Los Angeles, Los Angeles, California
  - Torrence Health Association, DBA Torrance Memorial;Physician Network/Cancer Care Associates, Redondo Beach, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Cancer Center of Santa Barbara with Sansum Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Rocky Mountain Cancer Centers - Denver Midtwon, Denver, Colorado
  - St. Mary's Hospital And Regional Medical Center, Grand Junction, Colorado
  - Memorial Healthcare System, Hollywood, Florida
  - Florida Cancer Affiliates, Ocala, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Florida Cancer Specialists & Research Institute, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Illinois Cancer Specialists, Niles, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Maryland Oncology Hematology P.A., Columbia, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - HCA Midwest Healthcare, Kansas City, Missouri
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Texas Oncology-Austin Central, Las Vegas, Nevada
  - Saint Barnabas Medical Cancer Center, Livingston, New Jersey
  - USOR - New York Oncology Hematology, P.C., Albany, New York
  - Hematology Oncology Associates, PC, Medford, Oregon
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Greenville Health System, Greenville, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, Lebanon, Tennessee
  - Texas Oncology - Baylor Charles A. Simmons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center-merge, Houston, Texas
  - Texas Oncology, P.A., San Antonio, Texas
  - Texas Oncology The Woodlands, The Woodlands, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Virginia Cancer Care Specialist, PC, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Wytheville, Virginia
- Germany (6):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Dresden
  - Local Institution, Essen
  - Local Institution, Freiburg im Breisgau
  - Klinikum Rechts der Isar der Technischen Universitaet Muenchen, München

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 239 participants were treated.
Groups:
- Advanced Malignancies Cohort: Treatment period 1: Nivolumab 240 mg Q2W for 8 doses. Treatment period 2: Nivolumab 480 mg Q4W
Period: Treatment Period 1
Arm/Group | Advanced Malignancies Cohort
Started | 239
Completed | 110
Not Completed | 129
Not completed — Disease progression | 90
Not completed — Adverse event unrelated to study drug | 12
Not completed — Death | 2
Not completed — Study Drug Toxicity | 6
Not completed — Participant request to discontinue | 9
Not completed — No longer meet study criteria | 1
Not completed — Participant withdrew consent | 3
Not completed — Other reasons | 6
Period: Transition From Period 1 to Period 2
Arm/Group | Advanced Malignancies Cohort
Started | 110
Completed (Completed = moved to Treatment Period 2) | 103
Not Completed | 7
Not completed — Other reasons | 1
Not completed — Participant withdrew consent | 1
Not completed — Death | 2
Not completed — Lost to Follow-up | 3
Period: Treatment Period 2
Arm/Group | Advanced Malignancies Cohort
Started | 103
Completed | 19
Not Completed | 84
Not completed — Disease progression | 69
Not completed — Adverse event unrelated to study drug | 1
Not completed — Maximum clinical benefit | 1
Not completed — Study Drug Toxicity | 5
Not completed — Participant request to discontinue | 2
Not completed — Participant withdrew consent | 3
Not completed — Other reasons | 3

BASELINE CHARACTERISTICS:
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 158
  Unknown or Not Reported | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 203
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR). Best overall response is defined as the best response designation, as determined by investigator, recorded in the specified timeframe, according to the RECIST 1.1 criteria.
Time Frame: From first dose to the date of objectively documented progression (per tumor-specific response criteria) or the date of subsequent therapy, whichever occurs first (up to approximately 24 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Percent of Participants | 7.9 [4.9 to 12.1]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first confirmed response (Complete Response, CR or Partial Response, PR) to the date of the first documented tumor progression (as determined by investigator) or death due to any cause, whichever occurs first.
  Median DOR computed using Kaplan-Meier method
Time Frame: From the time of first confirmed response to the date of the first documented progression (up to approximately 22 months)
Population: All Responders (Participants with a confirmed CR or PR)
Measure: Median (Full Range); unit: Months
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 19
Months | 21.78 [2.8 to 22.3]

3. Secondary Outcome: Time to Objective Response (TTR)
Description: TTR is defined as the time from first dosing date to the date of the first confirmed response (Complete Response, CR or Partial Response, PR), as assessed by investigator.
Time Frame: From the first dosing date to the date of the first confirmed response (up to approximately 10 months)
Population: All Responders (Participants with a confirmed CR or PR)
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 19
Months | 3.54 (2.337)

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with a best overall response of confirmed Complete Response (CR) or Partial Response (PR) or Stable Disease (SD).
Time Frame: From the first dosing date to the date of the last dose (approximately 24 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Percent of participants | 49.8 [43.3 to 56.3]

5. Secondary Outcome: Overall Survival Rate at 1 Year
Description: Overall Survival (OS) is defined as the time from the first dosing date to the date of death. A participant who has not died will be censored at last known date alive. OS rate at 1 year is measured as the percent of participants still alive at 1 year after first dosing, measured from Kaplan-Meier curve of OS.
Time Frame: From the first dosing date to 1 year later
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Percent of participants | 56.1 [49.1 to 62.5]

6. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died for any cause
Time Frame: From first dose to 100 days following last dose (up approximately 27 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Participants | 72

7. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Number of participants who experienced any grade, any cause AEs
Time Frame: From first dose to 30 days following the last dose (up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Participants | 234

8. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: Number of participants who experienced any grade, any cause SAEs
Time Frame: From first dose to 100 days following the last dose (up to approximately 27 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Participants | 148

9. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: Number of participants who experienced AEs leading to discontinuation of study therapy
Time Frame: From first dose to 30 days following the last dose (up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Participants | 41

10. Secondary Outcome: Number of Participants Experiencing Immune-mediated Adverse Events (IMAEs)
Description: Number of participants who experienced IMAEs. IMAEs are AEs consistent with an immune-mediated mechanism or immune-mediated component for which non-inflammatory etiologies (eg, infection or tumor progression) have been ruled out. IMAEs can include events with an alternate etiology which were exacerbated by the induction of autoimmunity.
Time Frame: From first dose to 100 days following the last dose (up to approximately 27 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Participants | 8

11. Secondary Outcome: Number of Participants Experiencing Select Adverse Events
Description: Number of participants who experienced Select Adverse Events. Select Adverse Events categories include: gastrointestinal, hepatic, pulmonary, renal, skin, hypersensitivity/infusion reaction.
Time Frame: From first dose to 30 days following the last dose (up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Participants
  Gastrointestinal Select AEs | 57
  Hepatic Select AEs | 33
  Pulmonary Select AEs | 6
  Renal Select AEs | 22
  Skin Select AEs | 59
  Hypersensitivity/Infusion Reaction | 7

12. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Dose Delay or Dose Reduction
Description: Number of participants who experienced AEs leading to dose delay or dose reduction. A dose will be considered as delayed if the delay is exceeding 3 days after the intended dose date (i.e., greater than or equal to 4 days from scheduled dosing date)
Time Frame: From first dose to 30 days following the last dose (up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 239
Participants | 61

13. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Specific Liver Tests
Description: Number of participants who experienced the laboratory abnormalities in specific liver tests described in the individual categories.
  ALT = Alanine Aminotransferase AST = Aspartate Aminotransferase ULN = Upper Limit of Normal
Time Frame: From first dose to 30 days following the last dose (up to approximately 25 months)
Population: All treated participants with available measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 231
Participants
  ALT OR AST > 3XULN | 11
  ALT OR AST > 5XULN | 8
  ALT OR AST > 10XULN | 3
  ALT OR AST > 20XULN | 1
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 230
  TOTAL BILIRUBIN > 2XULN | 5
  ALT OR AST > 3XULN + BILIRUBIN > 2XULN WITHIN 1 DAY: number analyzed (Participants) | 230
  ALT OR AST > 3XULN + BILIRUBIN > 2XULN WITHIN 1 DAY | 3
  ALT OR AST > 3XULN + BILIRUBIN > 2XULN WITHIN 30 DAYS: number analyzed (Participants) | 230
  ALT OR AST > 3XULN + BILIRUBIN > 2XULN WITHIN 30 DAYS | 3

14. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Specific Thyroid Tests
Description: Number of participants who experienced the laboratory abnormalities in specific thyroid tests described in the individual categories.
  TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal
Time Frame: From first dose to 100 days following the last dose (up to approximately 27 months)
Population: All treated participants with available measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Malignancies Cohort
Number analyzed (Participants) | 238
Participants
  TSH > ULN | 62
  TSH > ULN WITH TSH <= ULN AT BASELINE | 42
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 12
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUE >= LLN | 0
  TSH > ULN WITH FT3/FT4 MISSING | 2
  TSH < LLN | 38
  TSH < LLN WITH TSH >= LLN AT BASELINE | 25
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 8
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 1
  TSH < LLN WITH FT3/FT4 TEST MISSING | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion date (approximately 64 months). SAEs and Other AEs were assessed from first dose to 100 days following administration of the last dose (approximately 27 months).
Arm/Group | Advanced Malignancies Cohort
All-Cause Mortality (participants affected / at risk) | 156/239
Serious Adverse Events (participants affected / at risk) | 148/239
Other Adverse Events (participants affected / at risk) | 216/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Malignancies Cohort (N=239)
Anaemia (Blood and lymphatic system disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypophysitis (Endocrine disorders) | 1
Eye pain (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 5
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 6
Subileus (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 4
Localised oedema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 2
Sudden death (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Hepatic lesion (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Cholecystitis infective (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Enterocolitis infectious (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Infectious pleural effusion (Infections and infestations) | 2
Intervertebral discitis (Infections and infestations) | 1
Pelvic abscess (Infections and infestations) | 1
Perinephric abscess (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Renal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 8
Septic shock (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 2
C-reactive protein increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of cornea (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 58
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Penis carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Brain oedema (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Facial paralysis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Intracranial mass (Nervous system disorders) | 1
Neuritis cranial (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Venous stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Malignancies Cohort (N=239)
Anaemia (Blood and lymphatic system disorders) | 41
Hypothyroidism (Endocrine disorders) | 21
Abdominal pain (Gastrointestinal disorders) | 33
Abdominal pain upper (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 50
Diarrhoea (Gastrointestinal disorders) | 52
Dry mouth (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 53
Vomiting (Gastrointestinal disorders) | 32
Chills (General disorders) | 14
Fatigue (General disorders) | 90
Oedema peripheral (General disorders) | 24
Pyrexia (General disorders) | 24
Upper respiratory tract infection (Infections and infestations) | 17
Urinary tract infection (Infections and infestations) | 22
Alanine aminotransferase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 18
Blood alkaline phosphatase increased (Investigations) | 12
Blood creatinine increased (Investigations) | 15
Weight decreased (Investigations) | 22
Decreased appetite (Metabolism and nutrition disorders) | 37
Dehydration (Metabolism and nutrition disorders) | 23
Hypokalaemia (Metabolism and nutrition disorders) | 18
Hyponatraemia (Metabolism and nutrition disorders) | 15
Hypophosphataemia (Metabolism and nutrition disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 34
Back pain (Musculoskeletal and connective tissue disorders) | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Dizziness (Nervous system disorders) | 15
Headache (Nervous system disorders) | 19
Anxiety (Psychiatric disorders) | 13
Insomnia (Psychiatric disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 43
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44
Dry skin (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 26
Rash (Skin and subcutaneous tissue disorders) | 20
Hypertension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT02832167/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT02832167/SAP_001.pdf